CLINICAL TRIAL: NCT03614260
Title: The RADIANCE II Pivotal Study: A Study of the ReCor Medical Paradise System in Stage II Hypertension
Acronym: RADIANCE-II
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ReCor Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RADIANCE II Study
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Hypertension; Vascular Diseases; Cardiovascular Diseases
Keywords: Denervation; Resistant Hypertension; Essential Hypertension; Uncontrolled Hypertension
MeSH Terms: conditions — Hypertension; Vascular Diseases; Cardiovascular Diseases; Essential Hypertension

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Renal Denervation (Experimental): Renal Angiogram and Renal Denervation (Paradise Renal Denervation System)
  Interventions: Device: Paradise Renal Denervation System
- Sham Control (Sham Comparator): Renal Angiogram
  Interventions: Procedure: Renal Angiogram

INTERVENTIONS:
Device: Paradise Renal Denervation System — Following renal angiogram according to standard procedures, subjects remain blinded and are immediately treated with the renal denervation procedure after randomization.
  Other Names: Renal Angiogram; Renal Denervation
  Arms: Renal Denervation
Procedure: Renal Angiogram — Following renal angiogram to standard procedures, subjects remain blinded and renal angiogram is considered the sham procedure.
  Arms: Sham Control

SUMMARY:
The objective of the RADIANCE II Pivotal study is to demonstrate the effectiveness and safety of the Paradise System in subjects with Stage 2 hypertension on 0-2 medications at the time of consent. Prior to randomization, subjects will be hypertensive in the absence of hypertension medication.

ELIGIBILITY:
Inclusion Criteria:

* Previously or currently prescribed antihypertensive therapy
* Average office BP ≥ 140/90 mmHg <180/120 mmHg while stable for at least 4 weeks on 0-2 classes of antihypertensive medication
* Documented daytime ABP ≥ 135/85 mmHg and < 170/105 mmHg after 4-week washout/run-in period

Exclusion Criteria:

* Lacks appropriate renal artery anatomy for treatment
* Known, uncorrected causes of secondary hypertension other than sleep apnea
* Type I diabetes mellitus or uncontrolled Type II diabetes
* eGFR of <40
* Brachial circumference ≥ 42 cm
* Any history of cerebrovascular event or severe cardiovascular event, or history of stable or unstable angina within 12 months prior to consent
* Repeat (>1) hospitalization for hypertensive crisis within 12 months prior to screening period, or any hospitalization for hypertensive crisis within 3 months prior to screening period
* Chronic oxygen support or mechanical ventilation other than nocturnal respiratory support for sleep apnea
* Primary pulmonary hypertension
* Night shift workers
* Pregnant, nursing or planning to become pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2018-12-14 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of Major Adverse Events (MAE) | From baseline to 30 days post-procedure
Change in average daytime ambulatory systolic BP | From baseline to 2 months post-procedure

SECONDARY OUTCOMES:
Change in average 24-hr ambulatory systolic BP | From baseline to 2 months post-procedure
Change in average office systolic BP | From baseline to 2 months post-procedure
Change in average home systolic BP | From baseline to 2 months post-procedure
Change in average daytime ambulatory diastolic BP | From baseline to 2 months post-procedure
Change in average 24-hr ambulatory diastolic BP | From baseline to 2 months post-procedure
Change in average office diastolic BP | From baseline to 2 months post-procedure
Change in average home diastolic BP | From baseline to 2 months post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Kirtane, MD, SM, Principal Investigator — Columbia University Medical Center/New York-Presbyterian Hospital and the Cardiovascular Research Foundation; Prof. Michel Azizi, MD, PhD, Principal Investigator — Professor of Vascular Medicine, Hypertension Dept. and Clinical Investigation Center, Hôpital Européen Georges Pompidou
Locations (47):
- United States (28):
  - Cardiology PC, Birmingham, Alabama
  - Cedars Sinai Medical Center, Los Angeles, California
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Stamford Hospital, Stamford, Connecticut
  - MedStar Washington, Washington D.C., District of Columbia
  - The Cardiac and Vascular Institute, Gainesville, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Southern Illinois University, Springfield, Illinois
  - Ochsner Heart and Vascular Institute, New Orleans, Louisiana
  - The Brigham and Women's Hospital, Boston, Massachusetts
  - Munson Medical Center, Traverse City, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Saint Luke's Health System, Kansas City, Missouri
  - Renown Regional Medical Center, Reno, Nevada
  - Deborah Heart & Lung Center, Browns Mills, New Jersey
  - Hackensack University, Hackensack, New Jersey
  - Columbia University Medical Center/NYPH, New York, New York
  - Northwell Health Inc., New York, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - The University of Tennessee Health Science Center, Memphis, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - University of Utah, Salt Lake City, Utah
  - Swedish Medical Center, Seattle, Washington
- Centre Hospitalier Universitaire Saint-Pierre, Brussels, Belgium
- France (3):
  - Hôpital Saint André, Bordeaux
  - CHRU de Lille, Lille
  - Hôpital Européen Georges-Pompidou (HEGP), Paris
- Germany (6):
  - University Clinic Erlangen, Erlangen
  - University Clinic of Saarland - Homburg, Homburg
  - Klinikum Karlsruhe GmbH, Karlsruhe
  - Klinikum Konstanz, Konstanz
  - Herzzentrum Leipzig GmbH, Leipzig
  - Sana Kliniken Lübeck GmbH, Lübeck
- University Hospital Galway, Galway, Ireland
- Erasmus Medical Center, Rotterdam, Netherlands
- Hôpitaux Universitaires Genève, Geneva, Switzerland
- United Kingdom (6):
  - The Cardiothoracic Centre Basildon University Hospital, Basildon, Essex
  - University Hospitals Dorset NHS Foundation Trust, Bournemouth
  - Kent & Canterbury Hospital, Canterbury
  - University Hospital Wales, Cardiff
  - St Bartholomew's Hospital, London
  - Freeman Hospital, Newcastle upon Tyne

REFERENCES:
- [Result] Azizi M, Saxena M, Wang Y, Jenkins JS, Devireddy C, Rader F, Fisher NDL, Schmieder RE, Mahfoud F, Lindsey J, Sanghvi K, Todoran TM, Pacella J, Flack J, Daemen J, Sharp ASP, Lurz P, Bloch MJ, Weber MA, Lobo MD, Basile J, Claude L, Reeve-Stoffer H, McClure CK, Kirtane AJ; RADIANCE II Investigators and Collaborators. Endovascular Ultrasound Renal Denervation to Treat Hypertension: The RADIANCE II Randomized Clinical Trial. JAMA. 2023 Feb 28;329(8):651-661. doi: 10.1001/jama.2023.0713. PMID 36853250
- [Derived] Azizi M, Sharp ASP, Fisher NDL, Weber MA, Lobo MD, Daemen J, Lurz P, Mahfoud F, Schmieder RE, Basile J, Bloch MJ, Saxena M, Wang Y, Sanghvi K, Jenkins JS, Devireddy C, Rader F, Gosse P, Claude L, Augustin DA, McClure CK, Kirtane AJ; RADIANCE Investigators. Patient-Level Pooled Analysis of Endovascular Ultrasound Renal Denervation or a Sham Procedure 6 Months After Medication Escalation: The RADIANCE Clinical Trial Program. Circulation. 2024 Mar 5;149(10):747-759. doi: 10.1161/CIRCULATIONAHA.123.066941. Epub 2023 Oct 26. PMID 37883784
- [Derived] Kirtane AJ, Sharp ASP, Mahfoud F, Fisher NDL, Schmieder RE, Daemen J, Lobo MD, Lurz P, Basile J, Bloch MJ, Weber MA, Saxena M, Wang Y, Sanghvi K, Jenkins JS, Devireddy C, Rader F, Gosse P, Sapoval M, Barman NC, Claude L, Augustin D, Thackeray L, Mullin CM, Azizi M; RADIANCE Investigators and Collaborators. Patient-Level Pooled Analysis of Ultrasound Renal Denervation in the Sham-Controlled RADIANCE II, RADIANCE-HTN SOLO, and RADIANCE-HTN TRIO Trials. JAMA Cardiol. 2023 May 1;8(5):464-473. doi: 10.1001/jamacardio.2023.0338. PMID 36853627